CLINICAL TRIAL: NCT04057040
Title: A Phase 2 Study of the Hepcidin Mimetic PTG-300 in Patients With Phlebotomy-Requiring Polycythemia Vera
Brief Title: Hepcidin Mimetic in Patients With Polycythemia Vera (REVIVE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTG-300-04
Record Dates: First submitted 2019-08-07; First posted 2019-08-14 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Polycythemia Vera
Keywords: polycythemia vera
MeSH Terms: conditions — Polycythemia Vera

STUDY DESIGN:
Intervention Model Description: Part 1:
  28 week open-label dose escalation phase in which each subject's dose of PTG-300 is titrated to achieve a hematocrit <45%.
  Part 2:
  12-week blinded randomized withdrawal phase. Subjects are randomized 1:1 to continue PTG-300 or to receive placebo.
  Part 3:
  Up to 3 year open label extension.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 1 open label, Part 2 blinded, Part 3 open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose finding PTG-300 (Part 1); PTG-300 (Part 2); Open label extension PTG-300 (Part 3) (Experimental)
  Interventions: Drug: PTG-300
- Dose finding PTG-300 (Part 1); Placebo (Part 2); Open label extension PTG-300 (Part 3) (Experimental)
  Interventions: Drug: PTG-300; Drug: Placebo

INTERVENTIONS:
Drug: PTG-300 — Active
Drug: Placebo — Placebo
  Arms: Dose finding PTG-300 (Part 1); Placebo (Part 2); Open label extension PTG-300 (Part 3)

SUMMARY:
This is a Phase 2 study with an open-label dose escalation phase followed by a blinded withdrawal phase and an open label extension. The study is designed to monitor the PTG-300 safety profile and to obtain preliminary evidence of efficacy of PTG-300 for the treatment of phlebotomy-requiring polycythemia vera.

DETAILED DESCRIPTION:
Phase 2 study in approximately sixty subjects previously diagnosed with Polycythemia Vera who require phlebotomy on a routine basis. There is a 28 week dose finding phase to identify a dose that maintains hematocrit <45%. Subjects who successfully complete the dose finding phase will be entered into a 12 week randomized withdrawal phase to confirm the response. Subsequently patients will enter into an up to 3 year open label extension to investigate long term safety.

ELIGIBILITY:
Main Inclusion Criteria: All subjects must meet ALL of the following inclusion criteria to be enrolled.

1. Male and female subjects aged 18 years or older.
2. Meet revised 2016 World Health Organization (WHO) criteria for the diagnosis of polycythemia vera.
3. Records of all phlebotomies performed for at least 28 weeks (preferably up to 52 weeks) before dosing are available.
4. Subjects who are not receiving cytoreductive therapy must have been discontinued from any prior cytoreductive therapy for at least 24 weeks before screening and have recovered from any adverse events due to cytoreductive therapy.
5. Subjects receiving cytoreductive therapy with hydroxyurea, interferon, or ruxolitinib must have received cytoreductive therapy for at least 24 weeks and be on a stable dose or have a decreasing dose (Medical Monitor approval required) for at least 8 weeks before dosing and with no planned change in dose.

Main Exclusion Criteria: Subjects must meet NONE of the following exclusion criteria to be enrolled:

1. Active or chronic bleeding within 4 weeks of screening.
2. Meets the criteria for post-PCV myelofibrosis as defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT).
3. Known primary or secondary immunodeficiency.
4. Any surgical procedure requiring general anesthesia within 1 month prior to screening or planned elective surgery during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Proportion of responders during the blinded randomized withdrawal period (Week 29 to Week 41). | 12 weeks
  A subject will be considered a responder during the blinded randomized withdrawal phase if hematocrit control is maintained without phlebotomy eligibility.
  "Phlebotomy eligibility" is defined as any one of the following criteria being met:
  * hematocrit ≥45% that was ≥3% higher than Week 29 pre-randomization hematocrit value, or
  * hematocrit >48%, or
  * an increase of ≥5% in hematocrit compared to Week 29 pre-randomization hematocrit value.

SECONDARY OUTCOMES:
Change in rate of phlebotomy events between Week 17 through Week 29 (inclusive; 12 weeks) compared to each subject's historical rate. | 12 weeks
Change in rate of phlebotomy events between Week 1 through Week 29 (inclusive; 28 weeks) compared to each subject's historical rate. | 28 weeks
Proportion of subjects achieving a response at Week 29, with response defined as having achieved the absence of "phlebotomy eligibility" during the efficacy evaluation phase beginning at Week 17 and continuing to Week 29. | 12 Weeks
  "Phlebotomy eligibility" in Part 1 is defined as a hematocrit ≥45% that was ≥3% higher than baseline level (defined as Part 1 pre-dose Day 1) or a hematocrit >48%.
Proportion of subjects with reduction in the rate of phlebotomy events beginning at the Week 17 visit and continuing to Week 29 (12 weeks) compared to each subject's historical rate. | 12 Weeks
  Time to "phlebotomy eligibility" from Week 29 to Week 41/End of Part 2.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (14):
  - Mayo Clinic - Mayo Clinic Hospital, Phoenix, Arizona
  - Marin Cancer Care, Greenbrae, California
  - Stanford University, Palo Alto, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas, Westwood, Kansas
  - Pontchartrain Cancer Care, Covington, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Mount Sinai, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical Center, New York, New York
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- India (2):
  - Sahyadri Super Specialty Hospital, Pune, Maharashtra
  - All India Institute of Medical Sciences, Rishikesh, Uttarakhand

REFERENCES:
- [Derived] Kremyanskaya M, Kuykendall AT, Pemmaraju N, Ritchie EK, Gotlib J, Gerds A, Palmer J, Pettit K, Nath UK, Yacoub A, Molina A, Saks SR, Modi NB, Valone FH, Khanna S, Gupta S, Verstovsek S, Ginzburg YZ, Hoffman R; REVIVE Trial Investigators. Rusfertide, a Hepcidin Mimetic, for Control of Erythrocytosis in Polycythemia Vera. N Engl J Med. 2024 Feb 22;390(8):723-735. doi: 10.1056/NEJMoa2308809. PMID 38381675